CLINICAL TRIAL: NCT00238511
Title: An Open-Label Follow-on Trial to Assess the Long-Term Safety and Efficacy of Oral SPM 927 in Subjects With Postherpetic Neuralgia (PHN)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP0690
Record Dates: First submitted 2005-10-11; First posted 2005-10-13 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2009-09

CONDITIONS: Postherpetic Neuralgia
MeSH Terms: conditions — Neuralgia, Postherpetic | interventions — 2-(acetylamino)-3-methoxy-N-(phenylmethyl)-, (2R)-

INTERVENTIONS:
Drug: SPM 927

SUMMARY:
This trial was the follow-on trial to a preceeding double-blind, placebo controlled trial which included patients with at least moderate pain due to postherpetic neuralgia. It was conducted at six sites in Germany and has been clinically finalized. The patients had successfully completed the above mentioned trial in postherpetic neuralgia and, in the investigator's opinion, would benefit from long-term administration of Lacosamide. After a 1-week run-in phase the patients were uptitrated to their optimal dose and then continued into the maintenance phase. Dose adjustments were allowed throughout the trial.The change in pain was measured daily as well as interference of pain with sleep and general activity. As per protocol this trial was terminated after two years of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Postherpetic Neuralgia

Exclusion Criteria:

* Does not benefit from long term treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-11; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma
Locations (1):
- Schwarz, Monheim, Germany